CLINICAL TRIAL: NCT06079229
Title: Pilot Study of Geriatric Parameters and Quality of Life in Patients Over 70 Years Old Undergoing Pancreatic Cancer Surgery
Brief Title: Quality of Life in Elderly Patients After Pancreatic Cancer Surgery
Acronym: ADL_DPC_PA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0569; 2023-A01551-44 (Other: ID-RCB)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer; Surgery; Elderly
Keywords: Pancreatic cancer; pancreatectomy; pancreatic surgery; independence; quality of life; elderly people; octogenarian; geriatric assessment
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients over 70 undergoing pancreatic cancer surgery at the Édouard Herriot Hospital.: This is a non-comparative study, in which all subjects with histologically proven pancreatic cancer (all types) on biopsy or surgical specimen, operated on for this cancer (by cephalic duodenopancreatectomy or left pancreatectomy) at the Édouard Herriot Hospital since July 2021, aged 70 or older at the time of surgery, will be included in the same group.
  Interventions: Other: Phone call

INTERVENTIONS:
Other: Phone call — The only follow-up visit provided for in the protocol was a telephone contact 3 to 30 months after the patient's surgery. The rest of the data required for the study were obtained from the patient's medical records, collected in the course of routine practice.

SUMMARY:
Pancreatic cancer mainly affects the elderly, with over 85% of patients diagnosed after the age of 60 and over half after the age of 70. In France, the incidence of pancreatic cancer is currently around 14,000 new cases per year, making it the fourth leading cause of cancer death in women and the fifth in men.

Surgery is currently the only curative option available to patients, but it is not an option for many patients who already have metastatic or locally advanced cancer at the time of diagnosis. The main studies carried out on this type of intervention in the elderly focus on the surgical aspect, and the tolerability of such surgery is not well studied.

The aim of this study is to describe the impact of pancreatic surgery on the independence in daily activities and quality of life of patients aged over 70 with pancreatic cancer. These patients underwent surgery at Édouard Herriot Hospital (Hospices Civils de Lyon) since July 2021, and the assessment will be conducted through telephone questionnaires.

It is hypothesised that these patients will be able to maintain their independence in terms of daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically proven pancreatic cancer (all types) on biopsy or surgical specimen
* Operated on for this cancer (by cephalic duodenopancreatectomy or left pancreatectomy) at the Édouard Herriot Hospital since July 2021
* 70 years of age or older at the time of surgery.

Exclusion Criteria:

* Patients who have expressed their opposition to the study
* Patients under curatorship, guardianship or legal protection
* Patient unable to express non-opposition
* Patient unreachable after 4 attempted calls over 3 consecutive weeks
* Patient deceased at the time of the telephone call
* Persons deprived of their liberty by a judicial or administrative decision
* Persons under compulsory psychiatric care

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study focuses on adult patients over the age of 70 with pancreatic cancer (of any type) who have undergone pancreatectomy and have been operated on at the Édouard Herriot Hospital, Lyon, France since July 2021.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Evolution in the ADL questionnaire score between pre-operative and post-operative 3 to 30 months after surgery. | Between 3 months and 30 months after surgery.
  The ADL score (Activities of Daily Living) is designed to assess independence for activities of daily living. It is scored from 0 to 6, with 6 representing maximum independence for activities of daily living (washing, eating, dressing, etc.) and 0 a complete lack of independence.
  The significance of the difference in the ADL score before and after surgery will be tested using the Wilcoxon test.
  ADL will therefore be measured at 3 months after surgery at the earliest and at 30 months at the latest, at the time of the telephone call with the patient. The pre-operative value is recorded in the patient's file, measured a few weeks before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Byeul-A KIM, MD, Principal Investigator — Service de Gériatrie aigue, Hôpital Édouard Herriot, Hospices Civils de Lyon
Locations (1):
- Service de Gériatrie aigue, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon, France